CLINICAL TRIAL: NCT04291144
Title: Visualising the Cerebral Cholinergic Innervation and Parasympathetic Gastrointestinal Nerves in Patients With Dementia Lewy Bodies.
Brief Title: Visualising Cerebral and Peripheral Cholinergic Nerves in Patients With Dementia Lewy Bodies.
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: DLB-FEOBV
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-05

CONDITIONS: Dementia With Lewy Bodies; Degeneration Nerves; Positron-Emission Tomography; Acetylcholine
MeSH Terms: conditions — Lewy Body Disease; Nerve Degeneration | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Inclusion criteria are mild to moderate DLB, age above 50, ability to give informed consent.
  Interventions: Radiation: PET-CT using FEOBV; Radiation: MRI-scan; Diagnostic Test: Cognitive assessment; Diagnostic Test: Clinical assessment
- Healthy controls: Age above 50.
  Interventions: Radiation: PET-CT using FEOBV; Radiation: MRI-scan; Diagnostic Test: Cognitive assessment; Diagnostic Test: Clinical assessment

INTERVENTIONS:
Radiation: PET-CT using FEOBV — We will inject 300 MBq of 18F-FEOBV in a peripheral vein and scan the internal organs from (0-70 minutes). The patient then rests, and from 180-210min after injection, we will scan the brain on our Siemens High Resolution Research Tomograph.
Radiation: MRI-scan — All patients will have an MRI scan of the brain. T1-weighted images will be used to assess general anatomy and identify white matter. T2-weighted sequences will be performed to quantify competing brain pathology. Also, we will collect functional MRI data.
Diagnostic Test: Cognitive assessment — Full neuropsychometric examination including tests in 5 cognitive domains.
Diagnostic Test: Clinical assessment — Age, sex, duration of disease, patient history and full somatic and neurological examinations. Constipation assessed with Rome-III criteria. Evaluation of Rapid Eye Movement (REM) sleep Behaviour Disorder (RBDSQ) questionnaire. Test for orthostatic hypotension, heart rate variability, and deep breathing.

SUMMARY:
Lewy Body Dementia (DLB) is the second most common type of neurodegenerative dementia and characterized by loss of cholinergic neurons in the cerebrum and possibly also internal organs. A novel tracer, 18F-fluoroethoxybenzovesamicol (18F-FEOBV), binds to the cholinergic vesicle transporter, a protein expressed uniquely in the vesicles of cholinergic pre-synapses. Our aim is to investigate the cholinergic denervation in patients with DLB using 18F-FEOBV. The investigators plan to recruit 30 patients with DLB and 20 healthy controls to extensive cognitive assessment, computed and positron emission topography, magnetic resonance imaging, and samples of blood. The investigators hypothesize that patients with DLB, compared to controls, have decreased cholinergic innervation in cortical and subcortical areas of the brain, intestines and heart, and that the denervation corresponds to symptoms of autonomic and cognitive dysfunction.

DETAILED DESCRIPTION:
Dementia with Lewy Bodies (DLB) is the second most common type of neurodegenerative dementia after Alzheimer's disease. It is characterized by cognitive decline, cognitive fluctuations, visual hallucinations, parkinsonism, and sleep disturbances. There is evidence of cholinergic neuron loss in the cerebrum of DLB patients, and Lewy body pathology in the cholinergic parasympathetic nerves of internal organs. A novel tracer, 18F-fluoroethoxybenzovesamicol (18F-FEOBV), binds to the cholinergic vesicle transporter, a protein expressed uniquely in the vesicles of cholinergic pre-synapses, and therefore a very specific marker for cholinergic innervation. There is only one previous FEOBV publication in DLB (4 patients). That study showed impressive imaging quality, far better than earlier cholinergic PET-ligands, such as 11C-donepezil. Per Borghammer has pioneered the use of 11C-donepezil PET to visualize cholinergic loss, and 18F-FEOBV PET represents the next generation of high-resolution cholinergic imaging. The aim is to investigate the cholinergic denervation in patients with DLB using 18F-FEOBV. The investigators hypothesize that, compared to healthy elderly controls, patients with DLB show: (i) Cholinergic denervation in cortical and subcortical structures of the brain, and in peripheral organs, specifically the gut, pancreas, and heart. (ii) Correlations between cerebral cholinergic denervation and cognitive decline, assessed with neuropsychometric measures. (iii) Correlations between cholinergic denervation of internal organs and relevant symptoms of autonomic dysfunction, e.g. orthostatic hypotension and constipation, and with objective measures of autonomic malfunction, e.g. increased colonic transit time, increased intestinal volume, and reduced heart rate variability. (iv) Thinning of the vagal nerve detected by ultra sound. (v) Correlations between cerebral cholinergic denervation and perturbed neural networks measured by functional MRI. Secondary aims are to compare the cerebral uptake of 18F-FEOBV in DLB patients with/without markers of Alzheimer's Disease in the cerebrospinal fluid, relate the pattern of glucose uptake (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose, 18F-FDG PET) to that of 18F-FEOBV uptake in the cerebrum, and contribute to development of a diagnostic alpha-synuclein assay.

The investigators plan to include 25-30 DLB patients and 20 matched healthy elderly controls. Patients are recruited from the dementia clinic, Aarhus University. Inclusion criteria are mild to moderate DLB, ability to give informed consent, and typical signs of DLB on an 18F-FDG-PET scan. Exclusion criteria are major psychiatric, neurologic and medical comorbidities. The investigators will do a clinical assessment including full somatic and neurological examinations, an extensive neuropsychological cognitive assessment, assess autonomic symptoms and evaluate for sleep disorders, test for orthostatic hypotension and heart rate variability and colonic transit time. The investigators will inject 300 megabecquerel (MBq) of 18F-FEOBV in a peripheral vein and scan the internal organs from 0-70 minutes. The patient then rests, and from 180-210 minutes post-injection, the brain is imaged. This two-step method has been validated to give a robust estimate of the cholinergic innervation of the brain. The investigators will also do magnetic resonance imaging of the brain, ultrasound of vagal nerve, cerebrospinal fluid analysis and blood work. The investigators plan to write a manuscript describing the cerebral uptake of 18F-FEOBV as measure of cholinergic denervation of patients with DLB. A second manuscript will describe the uptake of 18F-FEOBV in the internal organs. A third manuscript will compare the cholinergic denervation of brain and organs to cognitive and autonomic symptoms. NO will participate in recruitment of patients, drafting of protocol and manuscripts, organizing logistics, analysis of data, and collecting clinical and paraclinical data. The investigators will pay particular attention the ethical issues of obtaining informed consent from demented persons and emphasize an evaluation of competence. The investigators expect that this method is better than the currently used 11C-donepezil, in which case it will replace its use for studies of cholinergic denervation in the future. Developing non-invasive PET imaging of short duration is particularly important in a demented patient population that often struggle to lie still during prolonged scanning sessions. Development of strong objective measures to aid diagnosis of DLB is important because DLB is a common disease projected to increase even further in prevalence in the years to come. Also, our side project of contributing to the development of a prion-assay to detect alpha-synuclein in the cerebrospinal fluid has promising clinical potential.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate DLB, ability to give informed consent, and typical signs of DLB on an FDG-PET or dopamine transporter (DaT)-scan

Exclusion Criteria:

* schizophrenia, bipolar disorder, cerebral neoplasms, clinical stroke, diabetes, peripheral neuropathy, previous surgery or radiotherapy on cerebrum or internal organs, gastrointestinal inflammatory disease, severe organ failure, allergy to CT-contrast media and contraindications to MRI-scans

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with DLB will be recruited from neurological and psychiatric departments in Denmark. Healthy controls will be recruited by advertising in local news papers.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Cerebral density of vesicular acetylcholine transporter in patients compared to controls | Day 1
  Average density will be determined in each group for relevant areas of the brain. Group differences will be calculated
Organ density of vesicular acetylcholine transporter in patients compared to controls | Day 1
  Average density will be determined in each group for intestine, pancreas, suprarenal gland, and heart. Group differences will be calculated
Density of vesicular acetylcholine transporter compared to cognitive profile and autonomic symptoms. | Day 2
  Obtain clinical information and perform standard neurologic and somatic evaluation and full neuropsychological assessment. Relate density of tracer in brain and organs to corresponding cognitive and autonomic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Per Borghammer, MD, DMSc, Study Chair — University of Aarhus
Locations (1):
- Department of Nuclear medicine and PET, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nejad-Davarani S, Koeppe RA, Albin RL, Frey KA, Muller MLTM, Bohnen NI. Quantification of brain cholinergic denervation in dementia with Lewy bodies using PET imaging with [18F]-FEOBV. Mol Psychiatry. 2019 Mar;24(3):322-327. doi: 10.1038/s41380-018-0130-5. Epub 2018 Aug 6. No abstract available. PMID 30082840